CLINICAL TRIAL: NCT02313142
Title: Responses of the Cardiovascular Systems to Leg Exercises in Microgravity-like Conditions
Acronym: STAMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Verena Klamroth, MD, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STAMAS_v1.1_Nov2014
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Deconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects (Experimental)
  Interventions: Behavioral: Leg exercises

INTERVENTIONS:
Behavioral: Leg exercises

SUMMARY:
One of the major issues in space explorations is the negative effect of prolonged exposure to very low gravity (i.e. a condition often referred to as microgravity or weightlessness) on astronauts' health. In this unusual condition the human body undergoes an adaptation process, often referred to as "deconditioning", that leads to significant loss of bone and muscle mass, hormonal changes, as well as modifications of important cardiovascular parameters. While the new physiological state is adequate to the microgravity environment, it results unsuitable upon return on earth. Hence after the mission astronauts experience various health-related problems and must undertake an intense rehabilitation program. Cardiovascular deconditioning originates mainly from a shift of blood from the lower extremities to the upper part of the body caused by the absence of gravity. In the long term (i.e. days) this causes a loss of blood and body fluid. In the short term (i.e. minutes) it elicits modifications to arterial blood pressure and heart rate.

In this study, funded by the European Union through the project STAMAS, we intend to evaluate whether leg physical exercises can lead to a displacement of blood towards the lower extremities, therefore ameliorating the upward fluid shift caused by weightlessness. More generally, we aim to investigate the short-term response of the cardiovascular system to leg exercises in microgravity-like conditions. After a clear understanding of these phenomena we will develop a controller that, by monitoring the physiological stare of a subject, will compute the appropriate exercise regime to stabilize his/her cardiovascular parameters to desired safe values. Our contribution will provide a better understanding of the cardiovascular system, and will delineate the physiological ground for the development of novel countermeasure devices against the cardiovascular deconditioning during space flight based on continuous leg exercises.

The protocol we propose in this document presents minimal risks for our potential subjects, while has the potential to produce important contributions. The cardiovascular parameters we intend to analyse are: blood pressure, heart rate and leg blood volume. These signals will be acquired non-invasively and with minimal risks. Leg exercises will be performed by means of a stepping device (MARCOS) previously developed in our Lab. MARCOS enables to vary the resistance applied against knee-extension movements, and therefore it allows a systematic evaluation of different exercise intensities. Finally, microgravity conditions can be easily emulated by letting the subjects lay on a tilted platform with head-down (i.e. head-down bed rest - HDBR, or head-down tilt - HDT) during the exercise sessions, thus inducing a shift of body fluid toward the thorax. The most effective inclination angle has proved to be as low as -6°, thus constituting only minimal risks for the subjects. In practice, subjects will comfortably lay on the negatively tilted platform and will perform stepping at different intensities while their cardiovascular parameters are being monitored and recorded in encrypted form for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Exclusion Criteria:

* Fracture lower extremities
* Restricted range of motion in hip, knee or ankle joint which restricts standing or walking
* Any injury limiting movements of the lower extremities
* Pregnancy
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc
* Presence of any psychiatric condition
* Tachycardia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Leg blood volume | 110 min

SECONDARY OUTCOMES:
Heart-rate | 110 min
Blood pressure | 110 min